CLINICAL TRIAL: NCT00350948
Title: Phase 3 Randomized Study of TLK286 (Telcyta®) in Combination With Liposomal Doxorubicin (Doxil/Caelyx)Versus Liposomal Doxorubicin (Doxil/Caelyx) as Second-Line Therapy in Platinum Refractory or Resistant Ovarian Cancer (ASSIST-5)
Brief Title: Phase 3 Randomized Study of Telcyta + Doxorubicin Versus Doxorubicin in Platinum Refractory or Resistant Ovarian Cancer
Acronym: ASSIST-5
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Telik (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLK286.3025
Record Dates: First submitted 2006-07-06; First posted 2006-07-11 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Ovarian Neoplasms
Keywords: Ovary
MeSH Terms: conditions — Ovarian Neoplasms | interventions — TER 286; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telcyta + Liposomal Doxorubicin (Experimental): Telcyta at 1000 mg/m2 followed by Liposomal Doxorubicin at 50 mg/m2 on Day 1 of each four-week treatment cycle
  Interventions: Drug: Telcyta; Drug: Liposomal Doxorubicin
- Liposomal Doxorubicin (Active Comparator): Liposomal Doxorubicin at 50 mg/m2 on Day 1 of each four-week treatment cycle
  Interventions: Drug: Liposomal Doxorubicin

INTERVENTIONS:
Drug: Telcyta — Day 1 of 28 day Cycle.
  Other Names: TLK286; canfosfamide
  Arms: Telcyta + Liposomal Doxorubicin
Drug: Liposomal Doxorubicin — Day 1 of 28 Day Cycle. 50 mg/m2
  Other Names: Doxil; Caelyx

SUMMARY:
The purpose of this research study is to determine if Telcyta® given in combination with liposomal doxorubicin is more effective than liposomal doxorubicin alone in treating women who have recurrent ovarian epithelial cancer, fallopian tube cancer or primary peritoneal cancer that is refractory or resistant to platinum chemotherapy.

DETAILED DESCRIPTION:
This is a randomized, open label, multicenter, multinational Phase 3 study of TLK286 (Telcyta) in combination with liposomal doxorubicin (Doxil/Caelyx) as compared to the active control therapy with liposomal doxorubicin (Doxil/Caelyx) as second line therapy in patients with platinum refractory or resistant recurrent ovarian cancer. Patients will be randomly assigned to receive either TLK286 (Telcyta) in combination with liposomal doxorubicin (Doxil/Caelyx) or active control liposomal doxorubicin (Doxil/Caelyx).

ELIGIBILITY:
Inclusion Criteria:

* Are a woman 18 years of age or older
* Have histologically or cytologically confirmed epithelial cancer or primary peritoneal cancer
* Have platinum refractory or resistant cancer
* Measurable disease according to radiographic RECIST criteria progression

Exclusion Criteria:

* Had treatment with first-line chemotherapy other than a platinum-containing regimen
* Have clinically significant cardiac disease
* Have any sign of intestinal obstruction interfering with nutrition
* Are pregnant or lactating
* Had prior treatment with liposomal doxorubicin
* Had prior treatment with Telcyta

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To demonstrate superiority in progression-free survival of TLK286 in combination with liposomal doxorubicin as compared with the active control arm liposomal doxorubicin | Once 244 planned pts. received at least 2 cycles of study treatment(s)

SECONDARY OUTCOMES:
To evaluate and compare the safety profile of each treatment arm | Any patient who received 1 dose of study treatment(s) will be evaluable for safety.

CONTACTS AND LOCATIONS:
Overall Officials: Gail L. Brown, MD, MBA, Study Director — Telik
Locations (71):
- United States (63):
  - Desert Oasis Cancer Center, Casa Grande, Arizona
  - Hematology Oncology Services of Arkansas, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - East Bay Medical Oncology/Hematology Medical Associates, Inc., Antioch, California
  - Bay Area Cancer Research Group, LLC, Concord, California
  - East Bay Medical Oncology/Hematology Medical Associates, Concord, California
  - California Oncology of the Central Valley, Fresno, California
  - Women's Cancer Research Foundation, Newport Beach, California
  - Southwest Cancer Care, Poway, California
  - Desert Hematology Oncology Medical Group, Rancho Mirage, California
  - Southern California Permanente Medical Group, San Diego, California
  - East Bay Medical Oncoogy/Hematology Medical Associates, Inc., San Leandro, California
  - Diablo Valley Oncology & Hematology Medical Group, Inc., Walnut Creek, California
  - Gynecologic Oncology Associates, Inc, Hollywood, Florida
  - Shands Jacksonville Medical Center, Jacksonville, Florida
  - University of Florida College of Medicine-Jacksonville, Jacksonville, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Florida Hospital, Orlando, Florida
  - Gynecologic Oncology Associates, Inc, Pembroke Pines, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Flossmoor Cancer Care (JOHA DBA), Flossmoor, Illinois
  - Joliet Oncology-Hematology Associates, Joliet, Illinois
  - Joliet Oncology-Hematology Associates, LTD., Joliet, Illinois
  - Kankakee Cancer Center (JOHA DBA), Kankakee, Illinois
  - Joliet Oncology-Hematology Associates, Morris, Illinois
  - St. Vincent Gynecologic Oncology, Indianapolis, Indiana
  - Central Baptist Hospital, Lexington, Kentucky
  - Hematology and Oncology Specialists, LLC, Metairie, Louisiana
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Arch Medical Services, St Louis, Missouri
  - Hematology & Oncology Consultants P.C., Omaha, Nebraska
  - Horizon's West Medical Group, Scottsbluff, Nebraska
  - The Women's Center of Western Nebraska, Scottsbluff, Nebraska
  - Schwaartz Gynecologic Oncology, PLLC, Babylon, New York
  - The Mary Imogene Bassett Hospital, Cooperstown, New York
  - Monter Cancer Center, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - Blumenthal Cancer Center, Charlotte, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Hospital, Charlotte, North Carolina
  - Piedmont Hematology Oncology Associates-Lexington Satellite, Lexington, North Carolina
  - Piedmont Hematology Oncology Associates, Winston-Salem, North Carolina
  - Dakota Cancer Institute/Dakota Clinic Ltd., Fargo, North Dakota
  - Gynecologic Oncology & Pelvic Surgery Associates, Columbus, Ohio
  - Garth Phibbs, M.D., FACOG, Toledo, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Kaiser Permanente NW, Oncology/Hematology, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Hematology & Oncology Associates of NEPA, Dunmore, Pennsylvania
  - Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania
  - Associates in Hematolog-Oncology, P.C., Upland, Pennsylvania
  - Carolina Center of Gynecologic Oncology, Charleston, South Carolina
  - Palmetto Health Alliance-Richland, Columbia, South Carolina
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Arlington Cancer Center, Arlington, Texas
  - Arlington Cancer Center, Trophy Club, Texas
  - Danville Hematology & Oncology, Inc., Danville, Virginia
  - Carilion GYN Oncology Associates, Roanoke, Virginia
- Belgium (3):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - A.Z. Groeninge Oncologish Centrum, Kortrijk
  - Universitaire Ziekenhuizen Leuven Dienst Oncologie, Leuven
- Brazil (3):
  - Hospital Vera Cruz-Instituto de Oncologia, Belo Horizonte, Minas Gerais
  - Centr de Oncologia do Instituto de Radiologia do Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, Cerqueria Cesar, São Paulo
  - Fundacao Hospital Amaral Carvalho, Rua Dona Siilveria, São Paulo
- United Kingdom (2):
  - Guy's & St. Thomas Cancer Centre, London, England
  - Ninewells Hospital and Medical School, Dundee, Scotland

REFERENCES:
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274
- [Derived] Vergote I, Finkler NJ, Hall JB, Melnyk O, Edwards RP, Jones M, Keck JG, Meng L, Brown GL, Rankin EM, Burke JJ, Boccia RV, Runowicz CD, Rose PG. Randomized phase III study of canfosfamide in combination with pegylated liposomal doxorubicin compared with pegylated liposomal doxorubicin alone in platinum-resistant ovarian cancer. Int J Gynecol Cancer. 2010 Jul;20(5):772-80. doi: 10.1111/igc.0b013e3181daaf59. PMID 20973267